CLINICAL TRIAL: NCT03466567
Title: A Trial Investigating the Effect of Probenecid and Ciclosporin on the Pharmacokinetics of SNAC in Healthy Subjects
Brief Title: A Trial Investigating the Effect of Probenecid and Ciclosporin on the Concentrations of SNAC in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4394; U1111-1197-9088 (Other: World Health Organization (WHO)); 2017-002498-21 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2018-03-09; First posted 2018-03-15 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide; Probenecid; Cyclosporine

STUDY DESIGN:
Intervention Model Description: This is a 3-period cross-over study. The participants will be randomised to three treatment sequences each consisting of three treatment periods. One treatment period with a single dose of 3 mg oral semaglutide alone, one treatment period with a single dose of 600 mg ciclosporin 1 hour prior to administration of a single dose of 3 mg oral semaglutide and one treatment period with 500 mg probenecid administered twice daily for 3½ days with the last dose 2 hours prior to administration of a single dose of 3 mg oral semaglutide. Pharmacokinetics of sodium N-(8-(2-hydroxybenzoyl) amino) caprylate (SNAC) and SNAC metabolites will be assessed after each single dose of 3 mg oral semaglutide.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Oral semaglutide, ciclosporin, probenecid (Experimental): Participants will receive oral semaglutide in treatment period 1, ciclosporin in treatment period 2, and probenecid in treatment period 3.
  Interventions: Drug: Semaglutide; Drug: Probenecid; Drug: Ciclosporin
- Probenecid, oral semaglutide, ciclosporin (Experimental): Participants will receive probenecid in treatment period 1, oral semaglutide in treatment period 2, and ciclosporin in treatment period 3.
  Interventions: Drug: Semaglutide; Drug: Probenecid; Drug: Ciclosporin
- Ciclosporin, probenecid, oral semaglutide (Experimental): Participants will receive ciclosporin in treatment period 1, probenecid in treatment period 2, and oral semaglutide in treatment period 3.
  Interventions: Drug: Semaglutide; Drug: Probenecid; Drug: Ciclosporin

INTERVENTIONS:
Drug: Semaglutide — A single dose of 3 mg semaglutide tablet alone will be administered orally. Trial product administration will take place in the morning after overnight fasting for at least 6 hours.
Drug: Probenecid — A dose of 500 mg probenecid (2 tablets of 250 mg) will be administered orally twice daily for 3½ days (7 trial product administrations in total). On the 4th day, the last probenecid administration will take place 2 hours prior to administration of a single dose of 3 mg oral semaglutide tablet. The last trial product administrations will take place in the morning after overnight fasting for at least 6 hours.
Drug: Ciclosporin — A single dose of 600 mg ciclosporin (6 capsules of 100 mg) will be administered orally 1 hour prior to administration of a single dose of 3 mg oral semaglutide tablet. Trial product administration will take place in the morning after overnight fasting for at least 6 hours.

SUMMARY:
The aim of the study is to investigate the effect of the medicines, probenecid and ciclosporin on the concentrations of SNAC. SNAC is an ingredient of the semaglutide tablets. Participants will get 3 different treatments (that is 3 treatment periods): 1) a single dose of 3 mg semaglutide, 2) a single dose of 600 mg ciclosporin with 3 mg semaglutide, 3) 500 mg probenecid twice a day for 3 ½ days with a single dose of 3 mg semaglutide on the last day.

The sequence of treatments participants get is decided by chance. Probenecid and ciclosporin are available medicines. They are given by doctors. Semaglutide contains SNAC. It cannot be prescribed yet.

The study will last for up to 125 days. Participants will have 17 to 18 visits at the study centre. This includes short visits at the centre for blood sampling only. Participants will have several blood draws.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of non-childbearing potential, aged 18-64 years (both inclusive) at the time of signing informed consent.
* Body mass index between 18.5 and 29.9 kg/sqm (both inclusive).
* Body weight greater than or equal to 50.0 kg.
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

- Use of tobacco and nicotine products, defined as: A. Smoking more than 1 cigarette or the equivalent per day B. Not able or willing to refrain from smoking and use of nicotine substitute products during the in-house period(s).

* Presence of clinically significant gastrointestinal disorders or symptoms of gastrointestinal disorders potentially affecting absorption of drugs or nutrients, as judged by the investigator.
* History (as declared by the subject) of major surgical procedures involving the stomach potentially affecting absorption of trial products (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery).
* Known glucose-6-phosphate-dehydrogenase deficiency (as declared by the subject).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

PRIMARY OUTCOMES:
AUC0-tz,SNAC,SD, area under the SNAC plasma concentration-time curve from time 0 to time of the last quantifiable concentration after a single dose of oral semaglutide | 0-48 hours
  Calculated based on plasma SNAC activity measured in blood.
Cmax,SNAC,SD, maximum observed SNAC plasma concentration on the concentration-time curve after a single dose of oral semaglutide | 0-48 hours
  Calculated based on plasma SNAC activity measured in blood.

SECONDARY OUTCOMES:
AUC0-tz,E494,SD, area under the SNAC metabolite E494 plasma concentration-time curve from time 0 to time of the last quantifiable concentration after a single dose of oral semaglutide | 0-48 hours
  Calculated based on plasma SNAC metabolite E494 activity measured in blood.
Cmax,E494,SD, maximum observed SNAC metabolite E494 plasma concentration on the concentration-time curve after a single dose of oral semaglutide | 0-48 hours
  Calculated based on plasma SNAC metabolite E494 activity measured in blood.
AUC0-tz,E506,SD, area under the SNAC metabolite E506 plasma concentration-time curve from time 0 to time of the last quantifiable concentration after a single dose of oral semaglutide | 0-48 hours
  Calculated based on plasma SNAC metabolite E506 activity measured in blood.
Cmax,E506,SD, maximum observed SNAC metabolite E506 plasma concentration on the concentration-time curve after a single dose of oral semaglutide | 0-48 hours
  Calculated based on plasma SNAC metabolite E506 activity measured in blood.
AUC0-∞,E1245,SD, area under the SNAC metabolite E1245 plasma concentration-time curve from time 0 to infinity after a single dose of oral semaglutide | 0-48 hours
  Calculated based on plasma SNAC metabolite E1245 activity measured in blood.
Cmax,E1245,SD, maximum observed SNAC metabolite E1245 plasma concentration on the concentration-time curve after a single dose of oral semaglutide | 0-48 hours
  Calculated based on plasma SNAC metabolite E1245 activity measured in blood.
AUC0-∞,E1246,SD, area under the SNAC metabolite E1246 plasma concentration-time curve from time 0 to infinity after a single dose of oral semaglutide | 0-48 hours
  Calculated based on plasma SNAC metabolite E1246 activity measured in blood.
Cmax,E1246,SD, maximum observed SNAC metabolite E1246 plasma concentration on the concentration-time curve after a single dose of oral semaglutide | 0-48 hours
  Calculated based on plasma SNAC metabolite E1246 activity measured in blood.
AUC0-∞,E1247,SD, area under the SNAC metabolite E1247 plasma concentration-time curve from time 0 to infinity after a single dose of oral semaglutide | 0-48 hours
  Calculated based on plasma SNAC metabolite E1247 activity measured in blood.
Cmax,E1247,SD, maximum observed SNAC metabolite E1247 plasma concentration on the concentration-time curve after a single dose of oral semaglutide | 0-48 hours
  Calculated based on plasma SNAC metabolite E1247 activity measured in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://www.novonordisk-trials.com/website/content/how-to-access-clinical-trial-datasets.aspx